CLINICAL TRIAL: NCT03980340
Title: Breath Biomarkers for Sleep Loss and Circadian Timing
Status: Terminated | Type: Observational
Why Stopped: Funding to carry out studies no longer available.
Sponsor: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Jeanne Duffy, Principal Investigator, Brigham and Women's Hospital
Other Study IDs: 2019-P-001628
Record Dates: First submitted 2019-05-23; First posted 2019-06-10 (Actual); Last update posted 2025-08-03 (Actual); Status verified 2025-07

CONDITIONS: Shift-Work Sleep Disorder; Shift Work Type Circadian Rhythm Sleep Disorder; Sleep Disorders, Circadian Rhythm; Sleep Disorders, Intrinsic; Advanced Sleep Phase Syndrome (ASPS); Advanced Sleep Phase Syndrome; Advanced Sleep Phase; Delayed Sleep Phase; Delayed Sleep Phase Syndrome; Non-24 Hour Sleep-Wake Disorder; Irregular Sleep-Wake Syndrome
Keywords: Sleep; Circadian Rhythms; Circadian Rhythm Disorder
MeSH Terms: conditions — Sleep Disorders, Circadian Rhythm; Sleep Disorders, Intrinsic; Chronobiology Disorders

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Saliva samples may be collected and assayed for cortisol.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: Short Nap Intervention — Study participants may be asked to have a 1-2 hour nap in between the breath analysis tests.
Behavioral: No Nap Intervention — Study participants may be asked to sit or lay down remaining awake for 1-2 hours in between breath analysis tests.

SUMMARY:
Insufficient sleep has both health and safety risks, but currently there are no quick, accurate and inexpensive ways to measure sleep deficiency. The current study aims to use a cutting-edge technology, small molecule analysis (e.g. metabolomics), to detect compounds in breath that reliably change with sleep-wake state and those whose levels vary by time of day.

DETAILED DESCRIPTION:
The goal of the study is to use a small molecule analysis (e.g. metabolomics) device to measure compounds in breath that may change with sleep-wake state and compounds that vary by time of day. Participants will be fitted with a plastic mask connected to the device for a breath analysis test for about 20 minutes. Then, participants may be asked to lie down and take a nap or to remain sitting/lying down for 1-2 hours. After such time, participants will be asked to complete another ~20 minute breath analysis test. Participants will be asked to complete questionnaires throughout the study session. Investigators may ask participants to provide up to two saliva samples during the study session. Participants will also be asked to complete a pre-study diary to document sleep/wake times, diet, and medications for the day before the study session. Participants may be asked if they would be willing to take part in an additional study session on another day.

ELIGIBILITY:
Inclusion Criteria:

* Healthy Adults who are able to fall asleep in the study conditions
* Beginning 2 hours before the study, participants will be asked to refrain from brushing their teeth, using mouthwash, eating or drinking anything (other than water), chewing gum, smoking, etc., until the study is complete.

Exclusion Criteria:

* Individuals on special diets (such as a very low carbohydrate diet) may be excluded
* Acute or debilitating medical condition
* Recent history of dental problems (gum disease, abcess, surgery) or current dental or mouth pain
* Current use of stimulants, hypnotics, tranquilizers, Central Nervous System active substances, and/or antibiotics.
* Use of products containing nicotine 24 hours prior to study

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Healthy volunteers will be recruited from the surrounding community.
Sampling Method: Non-Probability Sample
Enrollment: 5 (Actual)
Dates: Start 2021-01-28 (Actual); Primary Completion 2025-01-31 (Actual); Study Completion 2025-03-31 (Actual)

PRIMARY OUTCOMES:
Comparison of the change in composition of chemical analytes from the breath test | Study day 1
  The change in composition of chemical analytes from the breath analysis tests will be compared between the Short Nap Intervention and No Nap Intervention groups to see if there is a sleep-related change in the components of breath.
Change in composition of chemical analytes from the breath test | Study day 1
  The analytes present in individual subject's breath samples before and after a short nap (in the Short Nap Intervention) will be analyzed for differences in chemical composition.
Circadian differences in composition of chemical analytes from the breath test | Study day 1
  The analytes present in breath samples after a short nap (in the Short Nap Intervention) will be analyzed for differences in chemical composition depending on time of day (circadian variation).

CONTACTS AND LOCATIONS:
Overall Officials: Jeanne F Duffy, MBA, PhD, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States